CLINICAL TRIAL: NCT06554743
Title: Using Defaults to Reduce Harmful Environmental Impacts
Brief Title: Plant-Based Defaults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Chad Stecher@asu.edu, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00016889
Record Dates: First submitted 2024-07-29; First posted 2024-08-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Choice Behavior; Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Default Veg (Experimental): Received a plant-based meal as the default option on the event RSVP form that required participants to pre-select their meal choice
  Interventions: Behavioral: Default Veg
- Default Meat (Active Comparator): Received a meal with meat as the default option on the event RSVP form that required participants to pre-select their meal choice
  Interventions: Behavioral: Default Meat

INTERVENTIONS:
Behavioral: Default Veg — Received a plant-based meal as the default option on the event RSVP form that required participants to pre-select their meal choice
  Arms: Default Veg
Behavioral: Default Meat — Received a meal with meat as the default option on the event RSVP form that required participants to pre-select their meal choice
  Arms: Default Meat

SUMMARY:
In this study, participants at six different academic events were randomly assigned to one of two conditions: (1) a default meat group, where the default choice was a meal with meat and participants had the option of opting out and choosing a plant-based meal; and (2) a default veg group, where the default choice was a plant-based meal with the option of opting out and choosing a meal with meat. Based on the success of prior studies that implemented plant-based defaults through preselection, we hypothesized that more participants would choose the plant-based meal when that option was set as the default, and we hypothesized that the default intervention would be equally effective across academic institutions. We also hypothesized that the default intervention would be equally effective across demographic groups, which would help to further demonstrate the generalizability of our plant-based default intervention.

ELIGIBILITY:
Inclusion Criteria:

* Academic event attendee

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Proportion of participants selecting the plant-based meal | Immediately during the completion of the event RSVP form
  The percent (%) of participants selecting the plant-based meal option instead of the meal with meat option on the event RSVP from

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study will be share through the ASU Research Data Repository
Supporting Information: CSR, Analytic Code
Time Frame: Shortly after our manuscript is accepted for publication
Access Criteria: https://doi.org/10.48349/ASU/C1CWX9
URL: https://doi.org/10.48349/ASU/C1CWX9

REFERENCES:
- [Background] Zhang AW, Wharton C, Cloonan S, Boronowsky R, Magesh V, Braverman I, Marquez A, Leidy H, Wang MC, Cleveland DA, Jay J, Stecher C. Changing the default meal option at university events to reduce harmful environmental impacts: Six randomized controlled trials. Appetite. 2024 Sep 1;200:107572. doi: 10.1016/j.appet.2024.107572. Epub 2024 Jun 20. PMID 38908405